CLINICAL TRIAL: NCT03367871
Title: Phase II Single Arm Study of Combination Pembrolizumab, Chemotherapy and Bevacizumab in Patients With Recurrent, Persistent, or Metastatic Cervical Cancer
Brief Title: Combination Pembrolizumab, Chemotherapy and Bevacizumab in Patients With Cervical Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator left institution
Sponsor: University of Miami (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Abdulrahman Sinno, MD, Associate Professor of Clinical, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20170846
Record Dates: First submitted 2017-12-05; First posted 2017-12-11 (Actual); Results first posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-05

CONDITIONS: Cervical Cancer
Keywords: Recurrent Cervical Cancer; Persistent Cervical Cancer; Metastatic Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — pembrolizumab; Paclitaxel; Cisplatin; Carboplatin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab, Chemotherapy, Bevacizumab (Experimental): On day 1 of each 21 day cycle, participants will be administered Pembrolizumab 200mg (IV); Chemotherapy including Paclitaxel 175mg/m2 or 135 mg/m2 (IV), and Cisplatin 50mg/m2 (IV) or Carboplatin area under the curve (AUC) 5; and Bevacizumab 15mg/kg (IV).
  Interventions: Drug: Pembrolizumab; Drug: Paclitaxel; Drug: Cisplatin; Drug: Carboplatin; Drug: Bevacizumab

INTERVENTIONS:
Drug: Pembrolizumab — IV
  Other Names: MK-3475; Keytruda
Drug: Paclitaxel — Administered intravenously (IV) on day 1
  Other Names: Taxol
Drug: Cisplatin — Administered intravenously (IV) on day 1
  Other Names: Platinol
Drug: Carboplatin — Administered intravenously (IV) on day 1
  Other Names: Paraplatin
Drug: Bevacizumab — Administered intravenously (IV) on day 1
  Other Names: Avastin

SUMMARY:
The investigators propose to evaluate the efficacy of the combination of standard chemotherapy with bevacizumab with Pembrolizumab in women with recurrent, persistent, or metastatic cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed recurrent, persistent or metastatic (primary stage IVB) squamous cell carcinoma, adenosquamous carcinoma or adenocarcinoma of the cervix that is not amenable to curative treatment with surgery and/or radiation therapy.
2. All patients must have measurable disease as defined by Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.
3. Patients must have recovered from effects of recent surgery or radiotherapy or chemoradiotherapy.
4. Patients should be free of active infections requiring antibiotics (with the exception of uncomplicated urinary tract infection).
5. Tissue from an archival sample or newly obtained core or excisional biopsy of a tumor lesion within 6 weeks confirming diagnosis.
6. Age ≥ 18 years
7. Life expectancy > 3 months
8. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
9. Patients must have normal organ and marrow function as defined below:

   * Absolute neutrophil count (ANC) ≥1,500 /microliter (mcL)
   * Platelets ≥ 100,000 / mcL
   * Hemoglobin ≥ 8 g/dL or ≥ 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency
   * Serum creatinine ≤ 1.5 X upper limit of normal (ULN) OR Measured or calculated a creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≥ 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN. Creatinine clearance should be calculated per institutional standard.
   * Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
   * Aspartate transaminase (AST) (SGOT) and alanine transaminase (ALT) (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
   * Albumin ≥ 2.5 mg/dL
   * International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
   * Activated Partial Thromboplastin Time (aPTT) ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
10. Negative urine or serum pregnancy ≤72 hours (i.e. 3 days) prior to receiving the first dose of study medication if not surgically sterilized. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
11. Female subjects of childbearing potential (i.e., have not been surgically sterilized or have not been without menses for >1 year) should be willing to use 2 methods of birth control at the same time, be surgically sterile, or abstain from heterosexual activity for the course of the study and at least 120 days after the last study dose.
12. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer, are ineligible if there is any evidence of other malignancy being present within the last 5 years.
2. Patients who have had prior chemotherapy except when used concurrently with radiation therapy.
3. Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis other than for the treatment of cervical cancer within the last 5 years are excluded. Prior radiation for localized cancer of the breast, head and neck, or skin is permitted provided that it was completed more than 3 years prior to registration, and the patient remains free of recurrent or metastatic disease.
4. Patients with an ECOG performance status of 2, 3 or 4.
5. Has received prior therapy with an anti-programmed cell death protein 1 (PD-1), anti-PD-L1, or anti-PD-L2 agent.
6. Patients with known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
7. Patients with a known history of human immunodeficiency virus (HIV) or active bacillus tuberculosis (TB).
8. Known psychiatric or substance abuse disorders that would interfere with cooperation with requirements of the study
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (i.e., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. History of non-infectious pneumonitis that required steroids, evidence of interstitial lung disease or active, non-infectious pneumonitis, or history of pneumonitis requiring treatment.
11. Is pregnant, breastfeeding or expecting to conceive within the projected duration of the study, starting with the pre-screening or screening visit through 120 days after the last dose of study treatment.
12. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (HCV) (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
13. Received live vaccine within 30 days prior to the first dose of study treatment. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however. intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines and are not allowed.
14. Patient with known hypersensitivity to Pembrolizumab or any of its excipients (active ingredients).
15. Patient receiving concurrent additional biologic therapy.
16. Patients who are adults and unable to consent, who are not yet adults, pregnant and nursing women, and prisoners are ineligible.
17. Has an active infection requiring systemic therapy.
18. Thromboembolism (either arterial or venous) within 6 weeks of initiation of treatment.
19. Has significant cardiovascular disease, such as New York Heart Association cardiac disease classification of Class II or greater, myocardial infarction, or cerebrovascular accident within 3 months prior to initiation of study treatment, unstable arrhythmias, or unstable angina. Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or left ventricular ejection fraction <50% must be on a stable medical regimen that is optimized in the opinion of the treating physician in consultation with a cardiologist if appropriate.
20. Has undergone major surgical procedure within 28 days prior to first Bevacizumab dose or anticipation of the need for a major surgical procedure during the course of the study.
21. Has proteinuria, as demonstrated by urine dipstick or >2.0 g of protein in a urine protein-to creatinine ratio and/or 24 hour (hr) urine collection. All patients with ≥ 2+ protein on dipstick urinalysis at baseline must undergo a urine-to-protein ratio and/or 24 hr urine collection and demonstrate < 2.0 g of protein.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Huang, MD, MS, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab, Chemotherapy, Bevacizumab
Started | 17
Completed | 16
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab, Chemotherapy, Bevacizumab
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (OR)
Description: Objective response defined as the percentage of patients showing complete or partial response to study therapy. Response to therapy will be evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1).
Time Frame: Up to 24 months
Population: Participants who completed at least one cycle of study therapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab, Chemotherapy, Bevacizumab
Number analyzed (Participants) | 16
percentage of participants | 75 [53.8 to 96.2]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as percentage of participants without disease progression at time of study discontinuation will be assessed.
Time Frame: Up to 24 months
Population: Participants who received at least one dose of study therapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab, Chemotherapy, Bevacizumab
Number analyzed (Participants) | 17
percentage of participants | 48.7 [22.8 to 70.4]

3. Secondary Outcome: Overall Survival (OS)
Description: The rate of Overall Survival (OS) in study participants at 24 months will be reported. OS is defined as the time from the date of start of treatment until date of death due to any cause or date of last known to be alive. The estimate of OS rate at the 24 months is calculated by the Kaplan-Meier method, which takes into account the censored event-free times.
Time Frame: Up to 24 months
Population: Participants who received at least one dose of study therapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab, Chemotherapy, Bevacizumab
Number analyzed (Participants) | 17
percentage of participants | 58.3 [29.9 to 79.1]

4. Secondary Outcome: Number of Participants Experiencing Treatment-Related Toxicity
Description: The number of study participants experiencing treatment-related toxicity, including adverse events (AEs) and serious adverse events (SAEs), will be assessed. Treatment-related AEs and SAEs will be evaluated with respect to grade and relationship to treatment, using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 4.03.
Time Frame: Up to 15 months
Population: Participants who received at least one dose of study therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab, Chemotherapy, Bevacizumab
Number analyzed (Participants) | 17
Participants
  Treatment-related Serious Adverse Events (SAEs) | 2
  Treatment-related Adverse Events (AEs) | 14

ADVERSE EVENTS:
Time Frame: Up to 33 months.
Description: There were a total of seven deaths: Six patients died on study, one patient died off study.
Groups:
- Pembrolizumab, Chemotherapy, Bevacizumab: On day 1 of each 21 day cycle, participants will be administered Pembrolizumab 200mg (IV); Chemotherapy including Paclitaxel 175mg/m2 or 135 mg/m2 (IV), and Cisplatin 50mg/m2 (IV) or Carboplatin AUC 5; and Bevacizumab 15mg/kg (IV).
  Pembrolizumab: IV
  Paclitaxel: Administered intravenously (IV) on day 1
  Cisplatin: Administered intravenously (IV) on day 1
  Carboplatin: Administered intravenously (IV) on day 1
  Bevacizumab: Administered intravenously (IV) on day 1
Arm/Group | Pembrolizumab, Chemotherapy, Bevacizumab
All-Cause Mortality (participants affected / at risk) | 7/17
Serious Adverse Events (participants affected / at risk) | 6/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab, Chemotherapy, Bevacizumab (N=17)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Rectal Fistula (Gastrointestinal disorders) | 1 (1)
Anal Fistula (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) — Bacteremia
Urinary Tract Infection (Infections and infestations) | 2 (2)
Platelet count decreased (Investigations) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab, Chemotherapy, Bevacizumab (N=17)
Anemia (Blood and lymphatic system disorders) | 8 (11)
Myocarditis (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (2)
Hyperthyroidism (Endocrine disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 2 (2)
Blurred vision (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1) — Blepharitis
Watering eyes (Eye disorders) | 1 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1) — Rectal bleeding
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 4 (12)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) — Melena
Mucositis oral (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 4 (4)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (7)
Chills (General disorders) | 1 (1)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (3)
Fatigue (General disorders) | 11 (15)
Fever (General disorders) | 3 (3)
Infusion related reaction (General disorders) | 1 (2)
Localized edema (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 4 (5)
Vaginal infection (Infections and infestations) | 1 (1)
Vulval infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 8 (12)
Platelet count decreased (Investigations) | 1 (1) — Thrombocytopenia
Platelet count decreased (Investigations) | 2 (3)
Anorexia (Metabolism and nutrition disorders) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — Foot pain
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 3 (4)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 11 (14)
Restlessness (Psychiatric disorders) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (3)
Proteinuria (Renal and urinary disorders) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 1 (2)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Vaginal fistula (Reproductive system and breast disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — Discoloration skin, tongue
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 (3)
Hot flashes (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 7 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-22): https://cdn.clinicaltrials.gov/large-docs/71/NCT03367871/Prot_SAP_000.pdf